CLINICAL TRIAL: NCT00602030
Title: A Randomized, Placebo-controlled, Double-blind, Multicenter Phase 2 Study With a Lead in Phase of Erlotinib With or Without SNDX-275 in Patients With NSCLC After Failure In Up to Two Prior Chemotherapeutic Regimens for Advanced Disease
Brief Title: Study to Evaluate Erlotinib With or Without SNDX-275 (Entinostat) in the Treatment of Patients With Advanced NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SNDX-275-0401
Record Dates: First submitted 2008-01-25; First posted 2008-01-28 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Non-Small-Cell Lung Carcinoma; Carcinoma, Non-Small Cell Lung
Keywords: lung cancer; NSCLC; lung neoplasms; respiratory
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — entinostat; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Lead-in Phase: Erlotinib + Entinostat 5 mg (Experimental): Erlotinib 150 mg, tablets, orally, daily plus entinostat 5 mg, tablets, orally, on Days 1 and 15 of each 28-day cycle until disease progression or intolerable toxicities for up to 6 cycles in the Lead-in Phase.
  Interventions: Drug: Entinostat; Drug: Erlotinib
- Lead-in Phase: Erlotinib + Entinostat 10 mg (Experimental): Erlotinib 150 mg tablets, orally, daily plus entinostat 10 mg, tablets, orally, on Days 1 and 15 of each 28-day cycle until disease progression or intolerable toxicities for up to 6 cycles in the Lead-in Phase.
  Interventions: Drug: Entinostat; Drug: Erlotinib
- Double-blind Phase: Erlotinib + Entinostat 10 mg (Experimental): Erlotinib 150 mg, tablets, orally, daily plus entinostat 10 mg, tablets, orally, on Day 1 and 15 of a 28-day cycle until disease progression or intolerable toxicities for up to 6 cycles in the Double-blind Phase.
  Interventions: Drug: Entinostat; Drug: Erlotinib
- Double-blind Phase: Erlotinib + Placebo (Placebo Comparator): Erlotinib 150 mg, tablets, orally, daily plus placebo matching entinostat, tablets, orally, on Days 1 and 15 of each 28-day cycle until disease progression or intolerable toxicities for up to 6 cycles in the Double-blind Phase.
  Interventions: Drug: Placebo; Drug: Erlotinib
- Crossover Phase: Erlotinib + Entinostat 10 mg (Experimental): Participants in the Double-blind Phase Erlotinib + Placebo arm who experienced disease progression crossed over to receive open-label erlotinib 150 mg, tablets, orally, daily plus entinostat 10 mg, tablets, orally, on Days 1 and 15 of each 28-day cycle until disease progression or intolerable toxicities.
  Interventions: Drug: Entinostat; Drug: Erlotinib

INTERVENTIONS:
Drug: Entinostat — Entinostat tablets on Days 1 and 15 of a 28-day cycle.
  Other Names: SNDX-275
  Arms: Crossover Phase: Erlotinib + Entinostat 10 mg; Double-blind Phase: Erlotinib + Entinostat 10 mg; Lead-in Phase: Erlotinib + Entinostat 10 mg; Lead-in Phase: Erlotinib + Entinostat 5 mg
Drug: Placebo — Placebo-matching entinostat tablets on Days 1 and 15 of a 28-day cycle.
  Arms: Double-blind Phase: Erlotinib + Placebo
Drug: Erlotinib — Erlotinib 150 mg tablets once daily.
  Other Names: Tarceva

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of entinostat in combination with erlotinib in the treatment of Advanced Non-Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria

* Cytologically or histologically confirmed NSCLC of stage IIIb or IV
* Received at least 1 but no more than 2 prior chemotherapy or chemoradiotherapy regimens for advanced NSCLC (that did not include erlotinib and valproic acid) and progressed based on radiologic evidence
* At least 1 measurable lesion by conventional or spiral computed tomography (CT) scan
* Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1, or 2 and life expectancy of at least 6 months
* Paraffin-embedded tumor specimen available for correlative studies
* Male or female over 18 years of age
* Hemoglobin ≥ 9.0 g/dL; platelets ≥ 100 x 10^9/L; absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L without the use of hematopoietic growth factors
* Bilirubin and creatinine less than 2 times the upper limit of normal for the institution
* Albumin ≥ 2.5 g/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 3 times the upper limit of normal for the institution
* Prothrombin time less than 1.5 times the upper limit of normal for the institution
* Potassium, magnesium and phosphorus within the normal range for the institution (supplementation is permissible)
* Willing to use accepted and effective methods of contraception during the study (both men and women as appropriate) and for 3 months after the last dose of SNDX-275
* Patient or legally acceptable representative has granted written informed consent before any study-specific procedure (including special screening tests) are performed

Exclusion Criteria

* Prior stem cell transplant
* Clinical evidence of central nervous system (CNS) involvement
* Prior treatment with an histone deacetylase (HDAC) inhibitor or an epidermal growth factor receptor (EGFR) inhibitor
* Currently taking known inhibitors of CYPA4, including but not limited to atazanavir, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin, ≥ 10 mg prednisone, and voriconazole
* Currently taking medication(s) on the prohibited medication list
* Prior exposure to SNDX-275
* Systemic chemotherapy, radiotherapy, or treatment with an investigational agent without recovery to at least grade 1 or baseline before study drug administration
* Daily treatment with ≥ 10 mg prednisone within 28 days before study drug administration
* Local or whole brain palliative radiotherapy within 14 days before study drug administration
* Currently active second malignancy, or any malignancy within the last 5 years other than cured basal or squamous cell skin carcinoma, cervical carcinoma in situ, carcinoma in situ of the bladder, or papillary thyroid cancer
* Inability to swallow oral medications or a gastrointestinal malabsorption condition
* Acute infection requiring intravenous (IV) antibiotics, antivirals, or antifungals within 14 days before study drug administration
* Known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection
* Another serious or uncontrolled medical condition within 90 days before study drug administration such as acute myocardial infarction, angina, ventricular arrhythmias, hypertension, diabetes mellitus, or renal or hepatic insufficiency
* Known hypersensitivity to benzamides
* Women who are currently pregnant or breast-feeding
* Patient currently is enrolled in (or completed within 28 days before study drug administration) another investigational drug study
* Patient has any kind of medical, psychiatric, or behavioral disorder that places the patient at increased risk for study participation or compromises the ability of the patient to give written informed consent and/or to comply with study procedures and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2008-01-08 (Actual); Primary Completion 2010-02-04 (Actual); Study Completion 2012-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Witta, MD, Principal Investigator — Rocky Mountain Cancer Centers; Kartik Konduri, MD, Principal Investigator — Texas Oncology - Sammons Cancer Center; Robert Raju, MD, Principal Investigator — Dayton Oncology
Locations (30):
- United States (30):
  - HOPE (Hematology Oncology Physicians & Extenders), Tucson, Arizona
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Advanced Medical Specialties, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, Ocoee, Florida
  - Hematology Oncology Associates of Illinois, Chicago, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Kansas City Cancer Centers, Overland Park, Kansas
  - Alliance Hematology Oncology, Westminster, Maryland
  - St Joseph Oncology, Saint Joseph, Missouri
  - The Center for Cancer Care & Research, St Louis, Missouri
  - Mahonig Valley Hematology Oncology Associates, Boardman, Ohio
  - Dayton Oncology & Hematology, Kettering, Ohio
  - Oncology Associates of Oregon, Eugene, Oregon
  - Texas Oncology, Amarillo, Texas
  - Texas Oncology, Austin, Texas
  - Texas Oncology, Bedford, Texas
  - Texas Oncology, Sammons Cancer Center, Dallas, Texas
  - Texas Oncology, Dallas, Texas
  - Texas Oncology, Fort Worth, Texas
  - Texas Oncology, Garland, Texas
  - Texas Oncology, Longview, Texas
  - Texas Oncology, Midland, Texas
  - Texas Oncology, Odessa, Texas
  - Texas Oncology, Tyler, Texas
  - Fairfax Northern Virginia Hematology-Oncology, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Highline Medical Oncology, Burien, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 23 investigative sites in the United States from 8 January 2008 to 1 February 2012.
Pre-assignment Details: Participants with a diagnosis of non-small cell lung carcinoma (NSCLC) were enrolled in 5 or 10 mg entinostat plus erlotinib arms to determine the Phase 2 dose. Participants were enrolled 1:1 in treatment arms: erlotinib 150 mg + entinostat 10 mg or erlotinib 150 mg + placebo. Placebo arm could receive entinostat 10 mg in the Crossover Phase.
Period: Lead-in Phase
Arm/Group | Lead-in Phase: Erlotinib + Entinostat 5 mg | Lead-in Phase: Erlotinib + Entinostat 10 mg | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg | Crossover Phase: Erlotinib + Entinostat 10 mg
Started | 3 | 6 | 0 | 0 | 0
Completed | 1 | 1 | 0 | 0 | 0
Not Completed | 2 | 5 | 0 | 0 | 0
Not completed — Disease Progression | 2 | 3 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 0
Period: Double-blind Phase
Arm/Group | Lead-in Phase: Erlotinib + Entinostat 5 mg | Lead-in Phase: Erlotinib + Entinostat 10 mg | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg | Crossover Phase: Erlotinib + Entinostat 10 mg
Started | 0 | 0 | 65 | 67 | 0
Received Treatment | 0 | 0 | 63 | 65 | 0
Completed | 0 | 0 | 11 | 8 | 0
Not Completed | 0 | 0 | 54 | 59 | 0
Not completed — Disease progression | 0 | 0 | 33 | 30 | 0
Not completed — Adverse Event | 0 | 0 | 9 | 18 | 0
Not completed — Consent withdrawal | 0 | 0 | 4 | 3 | 0
Not completed — Death | 0 | 0 | 3 | 3 | 0
Not completed — Administrative decision | 0 | 0 | 0 | 2 | 0
Not completed — Ineligibility | 0 | 0 | 0 | 1 | 0
Not completed — Protocol deviation/noncompliance | 0 | 0 | 1 | 0 | 0
Not completed — Reason not specified | 0 | 0 | 4 | 2 | 0
Period: Crossover Phase
Arm/Group | Lead-in Phase: Erlotinib + Entinostat 5 mg | Lead-in Phase: Erlotinib + Entinostat 10 mg | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg | Crossover Phase: Erlotinib + Entinostat 10 mg
Started | 0 | 0 | 0 | 0 | 16
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 16
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3
Not completed — Consent withdrawal | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lead-in Phase: Erlotinib + Entinostat 5 mg | Lead-in Phase: Erlotinib + Entinostat 10 mg | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg | Total
Number analyzed (Participants) | 3 | 6 | 65 | 67 | 141
Age, Continuous [Median (Full Range); unit: years] | 72 [51 to 84] | 63.5 [46 to 78] | 67.0 [36 to 87] | 66.0 [32 to 90] | 67.1 [32 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 22 | 28 | 53
  Male | 2 | 4 | 43 | 39 | 88
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 6 | 55 | 55 | 119
  Black or African American | 0 | 0 | 6 | 5 | 11
  Asian | 0 | 0 | 2 | 1 | 3
  Hispanic | 0 | 0 | 1 | 6 | 7
  Other | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Identification of Safe-dose for the Phase 2 Double-blind Phase in the Lead-in Phase
Description: Safe recommended Phase 2 dose was determined based on dose-limiting toxicities (DLT) in Cycle 1. A DLT was defined as any of the following occurring in Cycle 1: Grade 3 or greater nonhematologic toxicity that was considered related to either entinostat or erlotinib or a Grade 4 hematologic toxicity lasting more than 7 days and/or resulting in a dose delay. Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 scale was used where Grade 1=mild, Grade 2=Moderate, Grade 3=Severe, medically significant, Grade 4=life-threatening and 5=death. The dose that was found to be safe is reported.
Time Frame: Cycle 1 of Lead-in Phase
Population: Lead-in Safety Analysis Set included all participant who received at least one dose of study drug in the Lead-in Phase.
Measure: Number; unit: milligrams (mg)
Groups:
- Lead-in Phase: Erlotinib + Entinostat: Participants received erlotinib 150 mg, tablets, orally, daily plus entinostat 5 mg or 10 mg, tablets, orally, on Days 1 and 15 of each 28-day cycle for up to 6 cycles in the Open-label Lead-in Phase 1 dose-finding study to identify a safe dose of entinostat in combination with erlotinib for further evaluation.
Arm/Group | Lead-in Phase: Erlotinib + Entinostat
Number analyzed (Participants) | 9
milligrams (mg) | 10

2. Primary Outcome: 4-Month Progression-free Survival (PFS) Rate in the Double-blind Phase
Description: PFS rate at 4 months was defined as the percentage of participants who are progression-free at 4 months.
Time Frame: Month 4
Population: Double-blind Per-protocol Analysis Set included all randomized participants who met key eligibility criteria, received an adequate course of treatment and who had baseline and postbaseline tumor measurements.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 50 | 53
percentage of participants | 24.0 [12.2 to 35.8] | 20.8 [9.8 to 31.7]
Statistical Analysis 1: Comparison: Double-blind Phase: Erlotinib + Placebo vs Double-blind Phase: Erlotinib + Entinostat 10 mg; Test type: Superiority; p = 0.505, Cochran-Mantel-Haenszel; Adjusted Odds Ratio = 0.72, 95% CI 2-sided [0.27 to 1.89] — Cochran-Mantel-Haenszel estimation of odds ratio adjusted for the smoking history stratification factor, using placebo as reference group

3. Secondary Outcome: Objective Response Rate (ORR) in the Double-blind Phase
Description: ORR was defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) as assessed by the investigator. CR=disappearance of all target lesions; disappearance of non-target lesions and normalization of tumor marker level. PR=At least a 30% decrease in the sum of the longest diameter of target lesions, taking at reference the baseline sum longest diameter.
Time Frame: Month 6
Population: Double-blind Full Analysis Set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 65 | 67
percentage of participants | 9.2 [2.2 to 16.3] | 3.0 [0.0 to 7.1]
Statistical Analysis 1: Comparison: Double-blind Phase: Erlotinib + Placebo vs Double-blind Phase: Erlotinib + Entinostat 10 mg; Test type: Superiority; p = 0.13, Cochran-Mantel-Haenszel; Adjusted Odds Ratio = 0.31, 95% CI 2-sided [0.06 to 1.54] — Estimation of odds ratio was adjusted for the smoking history stratification factor, using placebo as reference group

4. Secondary Outcome: 6-Month PFS Rate in the Double-blind Phase
Description: PFS rate at 6 months is defined as the percentage of participants who are progression-free at 6 months.
Time Frame: Month 6
Population: Full Analysis Set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 65 | 67
percentage of participants | 10.8 [3.2 to 18.3] | 11.9 [4.2 to 19.7]
Statistical Analysis 1: Comparison: Double-blind Phase: Erlotinib + Placebo vs Double-blind Phase: Erlotinib + Entinostat 10 mg; Test type: Superiority; p = 0.918, Cochran-Mantel-Haenszel; Adjusted Odds Ratio = 1.06, 95% CI 2-sided [0.34 to 3.27] — Estimation of odds ratio was adjusted for the smoking history stratification factor, using placebo as reference group

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) by Severity in the Double-blind Phase
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. Worsening of a pre-existing medical condition was considered an AE if there was either an increase in severity, frequency, or duration of the condition or an association with significantly worse outcomes. A TEAE is an AE that starts after the administration of study drug.
  A SAE is any AE that is fatal, life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth effect or other significant medical hazard.
  TEAE severity was graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 scale where Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, medically significant, Grade 4=Life-threatening and 5=Death.
Time Frame: First dose of study drug to within 30 days past last dose (Up to 7 months)
Population: Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 63 | 65
Participants
  Any SAE | 29 | 32
  Any TEAE | 63 | 65
  Grade 1 TEAE | 7 | 1
  Grade 2 TEAE | 16 | 12
  Grade 3 TEAE | 20 | 34
  Grade 4 TEAE | 5 | 6
  Grade 5 TEAE | 15 | 12

6. Secondary Outcome: Number of Participants With Grade 3 or 4 Laboratory Variables in the Double-blind Phase
Description: Laboratory tests included tests of Hematology and Chemistry. The individual laboratory values were graded by the investigator using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 scale where Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, medically significant, Grade 4=Life-threatening and 5=Death.
Time Frame: Day 1 and 15 of each cycle to safety follow-up 30 days past last dose (up to 7 months)
Population: Safety Population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 63 | 65
Participants
  White Blood Count decreased | 1 | 1
  Absolute Neutrophil Count decreased | 1 | 2
  Lymphocytes decreased | 9 | 18
  Platelets decreased | 1 | 2
  Phosphorus decreased | 4 | 6
  Alanine aminotransferase increased | 1 | 6
  Sodium decreased | 5 | 4
  Glucose increased | 2 | 3
  Albumin decreased | 4 | 2
  Potassium decreased | 2 | 2
  Aspartate aminotransferase increased | 0 | 2
  Bilirubin increased | 3 | 0
  Creatinine abnormal | 1 | 1
  Magnesium decreased | 0 | 1
  Potassium increased | 0 | 1
  Calcium increased | 2 | 0
  Calcium decreased | 1 | 0

7. Secondary Outcome: Vital Sign Values: Systolic Blood Pressure in the Double-blind Phase
Time Frame: Day 1 and 15 of each cycle to safety follow-up 30 days past last dose (up to 7 months)
Population: Safety Population included all participants who received at least one dose of study drug. Number analyzed is the number of participants with data available.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 63 | 65
mm Hg
  Baseline | 125.3 (17.41) | 126.0 (18.93)
  Minimum Post-Baseline Value: number analyzed (Participants) | 60 | 62
  Minimum Post-Baseline Value | 112.4 (13.95) | 105.0 (15.14)
  Maximum Post-Baseline Value: number analyzed (Participants) | 60 | 62
  Maximum Post-Baseline Value | 135.5 (15.74) | 132.5 (20.64)

8. Secondary Outcome: Vital Sign Values: Diastolic Blood Pressure in the Double-blind Phase
Time Frame: Day 1 and 15 of each cycle to safety follow-up 30 days past last dose (up to 7 months)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 63 | 65
mm Hg
  Baseline | 72.5 (10.06) | 72.1 (10.38)
  Minimum Post-Baseline Value: number analyzed (Participants) | 60 | 62
  Minimum Post-Baseline Value | 64.7 (9.31) | 61.3 (9.70)
  Maximum Post-Baseline Value: number analyzed (Participants) | 60 | 62
  Maximum Post-Baseline Value | 78.8 (9.92) | 78.5 (10.09)

9. Secondary Outcome: Vital Sign Values: Heart Rate in the Double-blind Phase
Time Frame: Day 1 and 15 of each cycle to safety follow-up 30 days past last dose (up to 7 months)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 63 | 65
beats per minute (bpm)
  Baseline | 87.5 (15.96) | 85.6 (17.41)
  Minimum Post-Baseline Value: number analyzed (Participants) | 60 | 62
  Minimum Post-Baseline Value | 78.5 (16.75) | 79.7 (15.19)
  Maximum Post-Baseline Value: number analyzed (Participants) | 60 | 62
  Maximum Post-Baseline Value | 98.2 (15.24) | 102.1 (17.12)

10. Secondary Outcome: Vital Sign Values: Respiration Rate in the Double-blind Phase
Time Frame: Day 1 and 15 of each cycle to safety follow-up 30 days past last dose (up to 7 months)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 63 | 65
breaths per minute
  Baseline: number analyzed (Participants) | 62 | 65
  Baseline | 18.5 (2.56) | 17.9 (2.46)
  Minimum Post-Baseline Value: number analyzed (Participants) | 60 | 62
  Minimum Post-Baseline Value | 17.2 (2.62) | 16.6 (2.34)
  Maximum Post-Baseline Value: number analyzed (Participants) | 60 | 62
  Maximum Post-Baseline Value | 20.2 (3.14) | 20.1 (2.66)

11. Secondary Outcome: Vital Sign Values: Temperature in the Double-blind Phase
Time Frame: Day 1 and 15 of each cycle to safety follow-up 30 days past last dose (up to 7 months)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: degrees Celsius (C)
Arm/Group | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 63 | 65
degrees Celsius (C)
  Baseline | 97.5 (0.84) | 97.6 (0.90)
  Minimum Post-Baseline Value: number analyzed (Participants) | 60 | 62
  Minimum Post-Baseline Value | 96.9 (1.15) | 97.0 (0.91)
  Maximum Post-Baseline Value: number analyzed (Participants) | 60 | 62
  Maximum Post-Baseline Value | 98.2 (0.90) | 98.5 (1.12)

12. Secondary Outcome: Vital Sign Values: Weight in the Double-blind Phase
Time Frame: Day 1 and 15 of each cycle to safety follow-up 30 days past last dose (up to 7 months)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 63 | 65
kilograms (kg)
  Baseline | 77.9 (16.83) | 74.3 (17.48)
  Minimum Post-Baseline Value: number analyzed (Participants) | 60 | 62
  Minimum Post-Baseline Value | 73.5 (16.98) | 70.0 (15.71)
  Maximum Post-Baseline Value: number analyzed (Participants) | 60 | 62
  Maximum Post-Baseline Value | 77.6 (16.97) | 74.3 (16.93)

13. Secondary Outcome: Cmax: Maximum Plasma Concentration of Entinostat in the Lead-in Phase
Time Frame: Day 1 predose and 0.5, 1, 2, 4 and 6 hours after dose; Days 2 and 8 predose (entinostat alone); Day 15 predose and 0.5, 1, 2, 4, 6 and 24 hours after dose
Population: Pharmacokinetic (PK) Population included all participants who had blood collected for PK parameters in the Lead-in Phase. Number analyzed is the number of participants with data available at the give timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lead-in Phase: Erlotinib + Entinostat 5 mg | Lead-in Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 3 | 6
ng/mL
  Day 1 (entinostat alone): number analyzed (Participants) | 3 | 5
  Day 1 (entinostat alone) | 19.6 (20.6) | 123.1 (136.4)
  Day 15 (entinostat + erlotinib): number analyzed (Participants) | 3 | 5
  Day 15 (entinostat + erlotinib) | 30.2 (41.0) | 99.4 (132.5)

14. Secondary Outcome: Tmax: Time to Cmax of Entinostat in the Lead-in Phase
Time Frame: as for outcome 13
Population: PK Population included all participants who had PK samples collected in the Lead-in Phase. Number analyzed is the number of participants with data available at the give time point.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Lead-in Phase: Erlotinib + Entinostat 5 mg | Lead-in Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 3 | 6
hour
  Day 1 (entinostat alone): number analyzed (Participants) | 3 | 5
  Day 1 (entinostat alone) | 0.83 (0.29) | 0.50 (0.00)
  Day 15 (entinostat + erlotinib): number analyzed (Participants) | 3 | 5
  Day 15 (entinostat + erlotinib) | 1.0 (0.9) | 1.3 (1.5)

15. Secondary Outcome: AUC(0-24): Area Under the Concentration-time Curve From Time 0 to 24 Hours in the Lead-in Phase
Time Frame: as for outcome 13
Population: PK Population included all participants who had PK samples collected in the Lead-in Phase. Number analyzed is the number of participants with data available at the given timepoint
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Lead-in Phase: Erlotinib + Entinostat 5 mg | Lead-in Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 3 | 6
ng*hr/mL
  Day 1 (entinostat alone): number analyzed (Participants) | 3 | 5
  Day 1 (entinostat alone) | 46.5 (12.2) | 133.3 (84.8)
  Day 15 (entinostat + erlotinib): number analyzed (Participants) | 3 | 5
  Day 15 (entinostat + erlotinib) | 51.7 (24.6) | 110.2 (92.3)

16. Secondary Outcome: AUC(0-last): Area Under the Concentration-time Curve From Time 0 to Last Quantifiable Concentration in the Lead-in Phase
Time Frame: as for outcome 13
Population: PK Population included all participants who had PK samples collected during the Lead-in Phase. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Lead-in Phase: Erlotinib + Entinostat 5 mg | Lead-in Phase: Erlotinib + Entinostat 10 mg
Number analyzed (Participants) | 3 | 6
ng*hr/mL
  Day 1 (entinostat alone): number analyzed (Participants) | 3 | 5
  Day 1 (entinostat alone) | 152.1 (26.3) | 325.8 (193.1)
  Day 15 (entinostat + erlotinib): number analyzed (Participants) | 3 | 5
  Day 15 (entinostat + erlotinib) | 51.7 (24.6) | 106.4 (96.8)

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days past last dose (up to 7 months)
Description: Number of participants at risk for Serious and Other Adverse events was based on the Safety Population that included all participants who received at least one dose of study drug.
Arm/Group | Lead-in Phase: Erlotinib + Entinostat 5 mg | Lead-in Phase: Erlotinib + Entinostat 10 mg | Double-blind Phase: Erlotinib + Placebo | Double-blind Phase: Erlotinib + Entinostat 10 mg | Crossover Phase: Erlotinib + Entinostat 10 mg
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/6 | 29/63 | 32/65 | 5/16
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 63/63 | 64/65 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-in Phase: Erlotinib + Entinostat 5 mg (N=3) | Lead-in Phase: Erlotinib + Entinostat 10 mg (N=6) | Double-blind Phase: Erlotinib + Placebo (N=63) | Double-blind Phase: Erlotinib + Entinostat 10 mg (N=65) | Crossover Phase: Erlotinib + Entinostat 10 mg (N=16)
Disease progression (General disorders) | 2 | 2 | 16 | 7 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Monoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (General disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 3 | 1
Anemia Group (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 1
Cardia disorder (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1 | 1 | 0
Dehydration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hernia obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia Group (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Superior vena caval occlusion (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Congestive cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-in Phase: Erlotinib + Entinostat 5 mg (N=3) | Lead-in Phase: Erlotinib + Entinostat 10 mg (N=6) | Double-blind Phase: Erlotinib + Placebo (N=63) | Double-blind Phase: Erlotinib + Entinostat 10 mg (N=65) | Crossover Phase: Erlotinib + Entinostat 10 mg (N=16)
Diarrhoea (Gastrointestinal disorders) | 1 | 6 | 30 | 37 | 3
Fatigue (General disorders) | 3 | 5 | 32 | 38 | 5
Nausea (Gastrointestinal disorders) | 1 | 3 | 16 | 32 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 35 | 33 | 1
Asthenia (General disorders) | 0 | 2 | 7 | 11 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 9 | 8 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 7 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 11 | 20 | 4
Oedema peripheral (General disorders) | 0 | 2 | 8 | 18 | 5
Thrombocytopenia group (Blood and lymphatic system disorders) | 0 | 2 | 2 | 10 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 7 | 11 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 8 | 20 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 6 | 2 | 0
Anemia group (Blood and lymphatic system disorders) | 2 | 1 | 7 | 15 | 3
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 10 | 26 | 2
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 6 | 9 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 4 | 5 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 4 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 7 | 6 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia group (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 4 | 1
Pyrexia (General disorders) | 0 | 1 | 5 | 4 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 6 | 9 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 6 | 3 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 2 | 8 | 0
Xerosis (General disorders) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 11 | 21 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 5 | 10 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 12 | 10 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 9 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 8 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 8 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 8 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 7 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 5 | 0
Depression (Psychiatric disorders) | 0 | 0 | 3 | 5 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 5 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 4 | 4 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 5 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 1 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Oedema (General disorders) | 0 | 0 | 0 | 0 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 3 | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 4 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 4 | 1
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results of the multi-center Study shall not be made before the first multi-site publication by Sponsor or Publications Committee. No Public Presentation by Institution or Investigator will be made until Study Documentation/Results from all sites are received and analyzed by Sponsor. Separate publication by Investigator will be delayed for a period of 18 months until the initial publication by Committee or Sponsor, or a determination is made not to make such publication.